CLINICAL TRIAL: NCT03223272
Title: Mechanisms of Refractory Hypertension (Reserpine)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Calhoun, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130822008
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Refractory Hypertension
Keywords: hypertension; sympathetic tone; resperpine
MeSH Terms: conditions — Hypertension | interventions — Reserpine

STUDY DESIGN:
Intervention Model Description: Open-label, dose titration study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reserpine (Experimental): Subjects will receive open-label reserpine 0.1 mg daily for 4 weeks.
  Interventions: Drug: Reserpine

INTERVENTIONS:
Drug: Reserpine — Open label reserpine 0.1 mg pill orally

SUMMARY:
The study is deigned to determine if refractory hypertension is attributable to heightened sympathetic tone by quantifying the antihypertensive benefit of reserpine, a sympatholytic agent, in patients failing other classes of antihypertensive agents.

DETAILED DESCRIPTION:
Patients with refractory hypertension, defined as uncontrolled office blood pressure despite use of 5 or more antihypertensive agents, including a thiazide diuretic and spironolactone. After withdrawal from other centrally-acting agents if needed, enrolled patients will be randomized to open-label reserpine 0.1 mg daily for 4 weeks. Twenty-four hour ambulatory blood pressure monitoring will be done at baseline, after the initial 4-week treatment period. All other antihypertensive medications will remain unchanged during the 4-week treatment period. The primary endpoint will be change in 24-hr ambulatory systolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

- adult with refractory hypertension defined as uncontrolled office blood pressure with use of 5 or more hypertensive agents, including a thiazide diuretic and spironolactone

Exclusion Criteria:

* congestive heart failure (EF 40%)
* chronic kidney disease (GFR <40 ml/min/1.73 mm)
* stroke and/or myocardial infarction or acute CHF exacerbation within last 3 months
* ongoing depression
* active peptic ulcer disease
* bradycardia <50 beats per minute
* 2nd or 3rd degree heart block
* known intolerance of reserpine
* use of digoxin or tricycle antidepressants

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Calhoun, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
One year after study completion, de-identified subject demographic data and primary outcome data will be available by request.
Supporting Information: Study Protocol
Time Frame: One year after study completion
Access Criteria: By request.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reserpine
Started | 7
Completed | 6
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Reserpine
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age +/- years
  years | 49.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Birmingham, AL, USA
  participants
    United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change Ambulatory Systolic Blood Pressure
Description: Twenty-four hour ambulatory systolic blood pressure
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Reserpine
Number analyzed (Participants) | 6
mmHg | -29.3 (22.2)

ADVERSE EVENTS:
Time Frame: Baseline through 10 weeks
Arm/Group | Reserpine
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reserpine (N=7)
NSTEMI (Cardiac disorders) | 1 (1) — Non ST-elevation MI

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT03223272/Prot_SAP_000.pdf